CLINICAL TRIAL: NCT07198152
Title: The Application of Artificial Intelligence in Screening Adrenal Nodules in Low-dose Chest CT
Brief Title: Artificial Intelligence Used in Screening Adrenal Nodules
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022yan068-002
Record Dates: First submitted 2025-08-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-09

CONDITIONS: Adrenal Incidentalomas; Thoracic CT-scan
Keywords: automatic segment; automatic classification
MeSH Terms: conditions — Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nodular adrenal glands: Adrenal region segmentation and adrenal nodule identification in chest CT via artificial intelligence
  Interventions: Other: None intervention
- Normal adrenal glands: Adrenal region delineation and adrenal gland identification in chest CT using artificial intelligence
  Interventions: Other: None intervention

INTERVENTIONS:
Other: None intervention — this study is retrospective based on the CT images, which dose include any intervention.

SUMMARY:
By collecting chest low-dose spiral CT plain scan images, extracting effective features from the adrenal gland regions, training and validating an artificial intelligence-based automatic diagnostic algorithm for adrenal nodules, we will ultimately develop an artificial intelligence software with independent intellectual property rights that is specifically designed for screening adrenal nodules in chest low-dose CT scans.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the population is over 18 years old, regardless of gender;
2. Images from chest low-dose CT plain scan during routine physical examination;

Exclusion Criteria:

1. Patients with a history of malignant tumors;
2. Imaging images with poor quality, artifacts, etc., which make analysis impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals aged over 18 years, with no gender restrictions, who underwent chest low-dose CT scans as part of routine physical examinations. Notably, those with a history of malignant tumors are excluded, and only individuals with qualified imaging data (free from poor quality, artifacts, or other issues that hinder analysis) are included.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Diagnostic Accuracy | From enrollment to the end of collection in one and a half years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MR-11-23-010450 — https://www.medicalresearch.org.cn